CLINICAL TRIAL: NCT01189214
Title: Psychopharmacotherapy in Multiple Substances Abuse / Dependence - the Pharmacological and Immunological Approach to the New Indication of Memantine
Brief Title: Psychopharmacotherapy in Multiple Substances Abuse
Acronym: MM opioid
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Opioid MM-2009; Taiwan NIH (Other Grant/Funding Number: DOH98-TD-I-111-DD004)
Record Dates: First submitted 2010-08-23; First posted 2010-08-26 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2010-08

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Memantine (Experimental)
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Add-on of memantine or placebo treatment will proceed in a double-blinded fashion for 12 weeks after adjusted methadone dose. During the study, we will evaluate treatment response and adverse effect from multiple dimensions to elucidate the therapeutic effect of add-on memantine on addictive behaviors. It will also explore the possible advantage of this treatment on social re-adaptation and psychopathogenesis of opioid dependence.

SUMMARY:
Add-on of memantine or placebo treatment will proceed in a double-blinded fashion for 12 weeks after adjusted methadone dose. During the study, the investigators will evaluate treatment response and adverse effect from multiple dimensions to elucidate the therapeutic effect of add-on memantine on addictive behaviors. It will also explore the possible advantage of this treatment on social re-adaptation and psychopathogenesis of opioid dependence.

DETAILED DESCRIPTION:
Opioid dependence is currently a severe problem for public health and social security. Methadone maintenance therapy may decrease the criminal rate and increase the quality of life for individuals with opioid dependence, but the high drop-out rate and long-term requirement to use of methadone are major problems in methadone maintenance therapy for opioid dependence. Methadone is after all another long acting opioid which may cause dependence. Therefore, current effort of methadone maintenance therapy is limited.

Memantine used to be recognized as a noncompetitive N-methyl-D-aspartate receptor antagonist. It was found with neuroprotective effects in several neurodegenerative diseases in recent few years. Memantine could inhibit brain inflammatory response through its action on reuroglial cells and provide neurotrophic effect. Previous studies also found memantine with inhibitory effects addictive behaviors in several substances. All of the above demonstrated that the combination of memantine and methadone in treating substance dependence prossess unique advantages, which may be superior to the original treatment. The main purpose of this study is to explore the neuroprotective effect of memantine on inhibition of brain inflammatory response through its action on reuroglial cells. Besides, we will evaluate the therapeutic effect of the combination of memantine and methadone in the subjects with opioid combine amphetamine dependence/abuse. It will also investigate multiple pathogenesis of addictive behaviors from the perspective of treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged ≧18 and ≦65 years.
2. A diagnosis of opioid abuse/dependence according to DSM-IV criteria made by a specialist in psychiatry.
3. A diagnosis of multiple drug abuse/dependence according to DSM-IV criteria made by a specialist in psychiatry.
4. Signed informed consent by patient or legal representative
5. Patient or a reliable caregiver can be expected to ensure acceptable compliance and visit attendance for the duration of the study.

Exclusion Criteria:

1. Women of childbearing potential not using adequate contraception as per investigator judgment or not willing to comply with contraception for duration of study.
2. Females who are pregnant or nursing.
3. Patients were diagnosed as other mental illness according to DMS-IV, except Major Depressive Disorder
4. Patient has received dextromethorphan, or other selective cyclo- oxygenase 2 (Cox-2) inhibitors, or other anti-inflammatory medication within 1 week prior to first dose of double-blind medication.
5. Current evidence of an uncontrolled and/or clinically significant medical condition (e.g., cardiac, hepatic and renal failure), which in the judgments of the investigator, would compromise patient safety or preclude study participation.
6. History of intolerance to valproate or memantine or other Cox-2 inhibitors.
7. History of sensitivity reaction (e.g., urticaria, angioedema, bronchospasm, severe rhinitis, anaphylactic shock) precipitated by memantine.
8. Patient has received electroconvulsive therapy (ECT) within 4 weeks prior to first dose of doubleblind medication.
9. Diagnosis of or treatment for esophageal, gastric, pyloric channel, or duodenal ulceration or related complications (bleeding and/or perforation) within 30 days prior to receiving first dose of double-blind medication.
10. Inclusion in another study of opioid dependence or study for another indication with psychotropic's within the last 30 days prior to start of study.
11. Increase in total SGOT, SGPT, BUN and creatinine by more than 3X ULN (upper limit of normal).
12. History of idiopathic or drug-induced agranulocytosis.
13. Substance-related disorders within 6 months prior to study start, borderline personality disorder, schizophrenia, or other major psychiatric disorders as defined by DSM-IV criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-03; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Urinary examination | baseline
  Using urinary examination is aimed to test whether the patient is using substance or not.
Urinary examination | week1
  Using urinary examination is aimed to test whether the patient is using substance or not.
Urinary examination | week2
  Using urinary examination is aimed to test whether the patient is using substance or not.
Urinary examination | week4
  Using urinary examination is aimed to test whether the patient is using substance or not.
Urinary examination | week8
  Using urinary examination is aimed to test whether the patient is using substance or not.
Urinary examination | week12
  Using urinary examination is aimed to test whether the patient is using substance or not.

SECONDARY OUTCOMES:
cytokines | baseline
cytokines | week1
cytokines | week2
cytokines | week4
cytokines | week8
cytokines | week12
lipid profiles | baseline, after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Band Lu, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- Ru-Band Lu, Tainan, Taiwan